CLINICAL TRIAL: NCT04704687
Title: Clinical Efficacy and Long Term Effects of Transcranial Direct Current Stimulation (tDCS) in Children With Attention Deficit/Hyperactivity Disorder (ADHD)
Acronym: STIMADHD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Hospices Civils de Lyon (Other); Nantes University Hospital (Other); Centre Hospitalier Charles Perrens, Bordeaux (Other Government); University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2018_843_0069
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Attention Deficit Hyperactivity Disorder; Transcranial Direct Current Stimulation
Keywords: Attention Deficit Hyperactivity Disorder; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tDCS (Experimental)
  Interventions: Other: Transcranial Direct Current Stimulation
- Sham (Active Comparator)
  Interventions: Other: Transcranial Direct Current Stimulation

INTERVENTIONS:
Other: Transcranial Direct Current Stimulation — Children will perform two successive interventions composed each by a set of 15 sessions of effective-tDCS combine with cognitive-training exercises.

SUMMARY:
Attention-Deficit/Hyperactivity Disorder (ADHD) is the most commonly diagnosed neurodevelopmental disorder in childhood. Patients with ADHD present inattention, impulsivity and hyperactivity causing severe impairments on academic achievement, social and professional life and daily functioning. Medications are effective in a majority of children with ADHD, but about 30% do not respond or tolerate stimulants, and some parents refuse pharmacological treatments.Transcranial Direct Current Stimulation is a safe and non-invasive technique of brain stimulation used in several neurological and psychiatric disorders, and recently in ADHD. In patients with ADHD, tDCS stimulations targeted frontal regions improve executive and attentional functioning and daily life symptoms. The objective of this project is to evaluate the efficacy of tDCS (vs sham) during cognitive-remediation exercises on ADHD symptoms (inattention, impulsivity and hyperactivity as defined by DSM-5) in children with ADHD between 7 and 14 years of age.

ELIGIBILITY:
* Children, male or females presenting a sufficient compliance for participate aged 7-14 years at the time of Visit 1 (Enrolment/baseline).
* Children's parent or legally authorised representative must sign informed consent. The children must sign assent if applicable (depending of age and understanding). The principal investigator of the center where the child is included signs the document, certifying that the family and the child, or their authorised representative, have received informed consents.
* Children meet DSM-5 criteria for ADHD (combined presentation) based on a clinical evaluation using questionnaire ADHD-Rating-Scale (ADHD-RS) and the Kiddie Schedule for Affective Disorders and Schizophrenia French version (Kiddie-SADS).
* Subjects have a minimum ADHD-RS total score of 32 at Visit 1.
* Children have a minimum CGI of 4 at Visit 1.
* Children have an age-appropriate intellectual level evaluated with WISC-5 (Full IQ >80).
* Children in which stimulant medication have been tested previously and stopped for adverse effects could be included in the study after a wash out of at least seven days.

Exclusion Criteria:

* Children have a neurological pathology or handicap: Epilepsy, cerebral palsy, sequelae of brain injury (traumatic or ischemic or inflammatory...)
* Children have a comorbid psychiatric disorder: conduct disorders, autism, severe obsessive-compulsive disorder, mood disorder, bipolar illness, conduct disorder, psychosis, and substance abuse.
* Children under medication (stimulant or other psychotropic treatment, benzodiazepine, antidepressant, hypnotics and melatonin) or who did not respond previously to stimulant will not be included.
* Severe sleep disorder.
* Contraindication to tDCS.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Variation of ADHD-RS(ADHD Rating Scale-IV) between both arms | at 4 weeks
  The ADHD Rating Scale-IV is completed independently by the parent and scored by a clinician. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. Results from this rating scale alone should not be used to make a diagnosis.
  How to Score
  For inattention (IA) subscale raw score: Add the odd-numbered items
  For hyperactivity-impulsivity (HI) subscale raw score: Add the even-numbered items
  To obtain the total raw score: Add the IA and Hi subscale raw scores
  Convert the raw scores to percentile scores by using the appropriate scoring profile provided on the back of the rating scale.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No